CLINICAL TRIAL: NCT06337630
Title: A Phase I Study on Tuvusertib (Oral ATR Inhibitor) in Combination With PLX038 (Topo1 Inhibitor) With Dose Expansion Cohorts in Patients With Advanced Solid Tumors
Brief Title: A Study on Tuvusertib (Oral ATR Inhibitor) in Combination With PLX038 (Topo1 Inhibitor) in Patients With Advanced Solid Tumors
Acronym: POP-ART
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Although no safety signal has been observed, given that the industrial development of tuvusertib has been halted regardless of the results, we see no scientific and ethical justification for continuing the study
Sponsor: Institut Curie (Other)
Collaborators: ProLynx LLC (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IC 2022-10
Record Dates: First submitted 2024-03-18; First posted 2024-03-29 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumor
Keywords: Pretreated; Metastatic; Locally; Advanced triple negative breast; ATM Gene Mutation
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: Phase I with a dose finding cohort, followed by expansion cohorts in pre-specified tumor types.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm: treatment with PLX038 and Tuvusertib (Experimental): Dose escalation step Dose escalation will be conducted on the grid defined by the 4 doses of PLX038 (800 mg/m², 1000 mg/m², 1300 mg/m² and 1700 mg/m² IV every 21 days D1=D22) and 3 doses of Tuvusertib (90 mg, 130 mg and 180 mg QD for 10 days from D3, D3-12). Premedication with anti-emetic agents is not required prior to the initial infusion, but may be used for an individual patient, as needed.
  Expansion cohorts Two expansion cohorts are planned, investigating the efficacy and safety in pre-specified populations of interest.
  Patients will be treated at the RP2D; 25 evaluable patients are needed in each cohort, to account for possible non evaluable patients, up to 28 patients will be enrolled in each cohort.
  Patients enrolled in the phase I part at the RP2D and fulfilling the eligibility criteria of one of the expansion cohorts will be counted in those 25 evaluable patients.
  Interventions: Drug: PLX038 + Tuvusertib

INTERVENTIONS:
Drug: PLX038 + Tuvusertib — Dose escalation will be conducted on the grid defined by the 4 doses of PLX038 (800 mg/m², 1000 mg/m², 1300 mg/m² and 1700 mg/m² IV every 21 days D1=D22) and 3 doses of Tuvusertib (90 mg, 130 mg and 180 mg QD for 10 days from D3, D3-12). Premedication with anti-emetic agents is not required prior to the initial infusion, but may be used for an individual patient, as needed.
  All included patients will receive PLX038 + Tuvusertib until progression of disease, unacceptable toxicity, patient withdrawal of consent, investigator decision, lost to follow-up, death, patient non-compliance, or study termination by Sponsor.

SUMMARY:
Phase I with a dose finding cohort, followed by expansion cohorts in pre-specified tumor types.

DETAILED DESCRIPTION:
This is an open label, multi-centric phase I with, first, a dose escalation step using an adaptation of the Bayesian Optimal INterval (BOIN) drug-combination, followed by 2 dose expansion cohorts using the Simon 2-stage design.

Dose escalation step Dose escalation will be conducted on the grid defined by the 4 doses of PLX038 (800 mg/m², 1000 mg/m², 1300 mg/m² and 1700 mg/m² IV every 21 days D1=D22) and 3 doses of Tuvusertib (90 mg, 130 mg and 180 mg QD for 10 days from D3, D3-12). Premedication with anti-emetic agents is not required prior to the initial infusion, but may be used for an individual patient, as needed.

starting combination level is c1 (PLX038 800mg/m2 and Tuvusertib 90mg). Groups of 3 patients will be sequentially enrolled. One week between the enrollment of the 1st patient and the 2 following patients is mandatory at a new combination level. The decision to (de)-escalate one of the two agents depends on the outcome of all patients treated at the current combination.

Expansion cohorts Two expansion cohorts are planned, investigating the efficacy and safety in pre-specified populations of interest.

Patients will be treated at the RP2D; 25 evaluable patients are needed in each cohort, to account for possible non evaluable patients, up to 28 patients will be enrolled in each cohort.

Patients enrolled in the phase I part at the RP2D and fulfilling the eligibility criteria of one of the expansion cohorts will be counted in those 25 evaluable patients.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to comply with the protocol and provide written informed consent prior to study-specific screening procedures.
* Age ≥ 18 years.
* Locally advanced or metastatic solid cancer that is not amenable to curative treatment.
* Measurable disease (per RECIST version 1.1).
* Received a minimum of one and a maximum of six prior cytotoxic chemotherapy regimens for locally advanced or metastatic cancer.
* Resolution of chemotherapy and radiation therapy related toxicities to NCI-CTCAE version 5.0 Grade 1 or lower severity, except for stable sensory neuropathy (≤ Grade 2), alopecia (any grade), presence of clinically managed chronic autoimmune AEs from prior immune therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate organ function (obtained within 14 days prior to treatment start) as evidenced by:

  i. Absolute neutrophil count (ANC) ≥ 1.5 X 109/L; ii. Hemoglobin (Hgb) ≥ 9 g/dL; iii. Platelet count ≥ 100 X 109/L; iv. Bilirubin ≤ 1.5 X upper limit of normal (ULN), except for patients with a documented history of Gilbert's disease (≤ 2 X ULN); v. Alanine aminotransferase (ALT), and aspartate aminotransferase (AST) ≤ 2.5 X ULN (for patients with liver metastases ≤ 5 X ULN); vi. Alkaline phosphatase (ALP) ≤ 3 X ULN (for patients with liver metastases, ≤ 5 X ULN); vii. Serum creatinine ≤ 1.5 mg/dL (133 μmol/L) or calculated creatinine clearance ≥ 50 mL/min (using Cockcroft-Gault formula); viii. Women of childbearing potential (WCBP): negative serum pregnancy test.
* Full blood count parameters described above must meet the thresholds with no transfusion or growth factor support in the past 14 days.
* Patients covered by social security or health insurance in compliance with the national legislation relating to biomedical research.
* The willingness to remain on contraception of childbearing potential for the duration of study treatment plus 7 months (women) or 4 months (men).

Exclusion Criteria:

* Patients who have had a last dose of IV chemotherapy within 21 days, last dose of oral cytotoxic chemotherapy, radiotherapy, biological therapy, or investigational therapy within 14 days prior to treatment start.
* Patients who have had any major surgery within 28 days prior to inclusion.
* Patients with chronic inflammatory bowel disease and/or bowel obstruction.
* Concomitant use of other agents for the treatment of cancer (except for LHRH agonist/antagonist) or any investigational agent(s).
* Brain metastases, unless local therapy was completed and use of corticosteroids for this indication discontinued for at least 3 weeks prior to inclusion. Signs or symptoms of brain metastases must be stable for at least 28 days prior to inclusion. No known progression of brain metastases (by imaging as assessed by RECIST version 1.1) can have occurred. Patients with leptomeningeal disease or meningeal carcinomatosis are excluded.
* Women who are either pregnant, lactating, planning to get pregnant.
* Patients receiving pharmacotherapy for hepatitis B or C, tuberculosis, or HIV.
* Patients with known liver disease diagnosed with Child-Pugh A or higher cirrhosis.
* Other current or previous stage III or IV malignancy diagnosed within 5 years of study entry.
* Severe/uncontrolled intercurrent illness within the previous 28 days prior to inclusion.
* Uncontrolled or poorly controlled arterial hypertension, symptomatic congestive heart failure (New York Heart Association Classification ≥ Class III), uncontrolled cardiac arrhythmia, calculated QTc average using the QTcF > 480 msec; unstable angina pectoris, myocardial infarction or a coronary revascularization procedure, cerebral vascular accident, transient ischemic attack, or any other significant vascular disease within 180 days of study intervention start.
* Patients with ongoing active infection (requiring systemic treatment) and treatment with live or live attenuated vaccine within 30 days of dosing.
* Any other significant medical, psychological, social or geographic conditions that in the opinion of the Investigator would impair study participation or cooperation.
* Patients deprived of their liberty or under guardianship.

Dose expansion additional inclusion criteria

Breast cancer

* Triple-negative breast cancer (both ER and PR <10%, HER2-negative or HER2-low, locally assessed).
* Prior therapy (administered in the neoadjuvant, adjuvant and/or metastatic setting) with an anthracycline, taxane and sacituzumab govitecan (unless not medically appropriate or contraindicated for the patient).
* Patients with known gBRCA mutations must have received a PARP inhibitor in the metastatic setting.
* Patients whose cancer has a CPS score ≥10 must have received prior pembrolizumab unless (i) contra-indicated (ii) CPS score or pembrolizumab not available at time of first line treatment start.

ATM-mutated solid cancers

● Inactivating mutation of ATM (presence of truncating mutation or R337/R3008 missense mutation of ATM mono and/or biallelic, assessed by next-generation sequencing in a certified French genomics platform).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2025-01-20 (Actual); Primary Completion 2025-11-24 (Actual); Study Completion 2025-11-24 (Actual)

PRIMARY OUTCOMES:
Dose escalation step : Dose limiting toxicities (DLTs) | 21 days
  Dose limiting toxicities (DLTs) experienced during 21 days from the first IV infusion of PLX038 + Tuvusertib
Expansion cohorts : Best tumor response | 6 months
  Best tumor response (defined as PR or CR in the first 6 months of treatment, assessed by investigators per RECIST v1.1 criteria)
Expansion cohorts : Serious Adverse Events (SAEs) | Until 30 days after the last dose of IMP (44 months + 30 days)
  Serious Adverse Events (SAEs) according to NCI CTCAE v5.0 by grade and their relationship to PLX038 + Tuvusertib.
Expansion cohorts : Adverse Events (AEs) | Until 30 days after the last dose of IMP (44 months + 30 days)
  Adverse Events (AEs) according to NCI CTCAE v5.0 by grade and their relationship to PLX038 + Tuvusertib.

SECONDARY OUTCOMES:
Dose escalation step : Pharmacokinetics effect of PLX038 and Tuvusertib | through study completion, an average of 44 months
  Maximum Plasma Concentration effect of PLX038, SN38 and Tuvusertib
Dose escalation step : Pharmacodynamics effect of PLX038 and Tuvusertib | through study completion, an average of 44 months
  Maximum Plasma Concentration effect of PLX038, SN38 and Tuvusertib
Dose escalation step : objective response rate (ORR) | through study completion, an average of 44 months
  ORR defined as the percentage of patients with complete response (CR) or partial response (PR), as the best response measured at the disease assessmement after initiation of treament according to RECIST v1.1
Dose escalation step : Time to response (TTR) | through study completion, an average of 44 months
  TTR calculated from the initiation of treatment to best tumour response (CR/PR)
Dose escalation step : Duration of Response (DoR) | through study completion, an average of 44 months
  DoR defined as the time period from best tumour response to disease progression (according to RECIST v1.1)
Dose escalation step : Progression free survival (PFS) | through study completion, an average of 44 months
  PFS measured from the inclusion in the study to the first documented progression (according to RECIST v1.1) or death from any cause.
Expansion cohorts : Time to response (TTR) | through study completion, an average of 44 months
  TTR calculated from the initiation of treatment to best tumour response (CR/PR)
Expansion cohorts : Duration of Response (DoR) | through study completion, an average of 44 months
  DoR defined as the time period from best tumour response to disease progression
Expansion cohorts : Progression free survival (PFS) | through study completion, an average of 44 months
  PFS measured from the inclusion in the study to the first documented progression
Expansion cohorts : Overall Survival (OS) | through study completion, an average of 44 months
  OS is defined as the time from inclusion to the event death.
Expansion cohorts : Efficacy of PLX038 + Tuvusertib in pre-defined biomarker subgroups | through study completion, an average of 44 months
  Association between PLX038 + Tuvusertib efficacy and homologous recombination (HR) defect (assessed by HR genes mutational status and BCRAness phenotype), replication stress-related biomarkers such as SFLN11 expression, RB1 loss; genomic alterations in DDR genes
Expansion cohorts : Pharmacokinetics effect of PLX038 and Tuvusertib | through study completion, an average of 44 months
  Maximum Plasma Concentration effect of PLX038, SN38 and Tuvusertib
Expansion cohorts : Pharmacodynamics effect of PLX038 and Tuvusertib | through study completion, an average of 44 months
  Maximum Plasma Concentration effect of PLX038, SN38 and Tuvusertib
Exploratory endpoints | through study completion, an average of 44 months
  Association between PLX038 + Tuvusertib efficacy and quantitative changes of blood biomarkers (e.g. ctDNA) during therapy.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Institut Curie, Paris
  - Institut Curie, Saint-Cloud

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets. Documents generated under the project will be disseminated in accordance with Institut Curie policies.
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).